CLINICAL TRIAL: NCT06895005
Title: Effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation on Upper Limb Motor Recovery After Stroke
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Patients With Stroke
Acronym: INPULSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Ministerio de Ciencia Tecnología e Innovación - Minciencias (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEI-2021-03209
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Motor Impairment; Motor Impairments; Stroke; Stroke; Sequelae; Stroke, Ischemic
Keywords: Stroke; Vagus nerve; Vagus nerve stimulation; Transcutaneous vagus nerve stimulation; Rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A double blinding will be performed. This information will be guaranteed to remain masked until after the analysis is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation + rehabilitation therapy (Experimental)
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation + rehabilitation therapy
- Sham stimulation + rehabilitation therapy (Sham Comparator)
  Interventions: Other: sham stimulation + rehabilitation therapy

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation + rehabilitation therapy — Transcutaneous auricular vagus nerve stimulation using INPULSE 3 times a week for six consecutive weeks. The stimulation parameters will be a frequency of 30Hz with a pulse width of 300 us and a stimulation time of 1.5 seconds for each respiratory cycle. The electrical current will be gradually increased to a maximum of 5 mA (0.25-mA increments) to allow adaptation to the stimulation until a comfortable tolerance level is achieved. Patients will receive physical rehabilitation therapy during stimulation, which will include reaching and grasping exercises, gross movements, turning objects, simulating specific tasks, inserting objects, opening and closing containers.
  Arms: Transcutaneous auricular vagus nerve stimulation + rehabilitation therapy
Other: sham stimulation + rehabilitation therapy — Patients will receive physical rehabilitation therapy during placebo stimulation (No electrical stimulation), including reaching and grasping exercises, gross movements, turning objects, simulating specific tasks, inserting objects, opening and closing containers.
  Arms: Sham stimulation + rehabilitation therapy

SUMMARY:
This study will evaluate the effects of transcutaneous vagus nerve stimulation in combination with physical rehabilitation on upper limb motor function of patients with stroke.

DETAILED DESCRIPTION:
Stroke is a neurological condition caused by vascular problems such as cerebral infarction and/or intracerebral or subarachnoid hemorrhage(1). In 2019, more than 12 million strokes occurred worldwide, making it one of the leading causes of morbidity.

Motor impairment is considered one of the main problems resulting from this condition(2). Recovery of motor function occurs spontaneously during the first months after stroke(3) as a result of brain plasticity processes in the sensory and motor systems(4). It is estimated that 50 to 75% of patients with stroke persist with significant motor sequelae limiting daily activities(5).

Recently, Vagus Nerve Stimulation (VNS) has been proposed as an intervention that could have beneficial effects in the recovery of motor function in these patients, since it contributes to the generation of adaptive neuroplasticity and the activation of neuromodulators that reduce brain inflammation(6).

VNS has mainly been administered by using implanted electrodes, but more recently, a non-invasive technique, known as transcutaneous VNS (cervical or auricular) has been proposed. VNS has traditionally required the implantation of an electrical pulse generator at the left subclavicular level, which is connected to electrodes in the left cervical branch of the vagus nerve(7). Its insertion is performed by a surgical procedure, which presents a higher risk of adverse events(8), the most frequent being dysphonia during stimulation, due to its proximity to the laryngeal nerve(9). On the other hand, transcutaneous VNS works through the placement of non-invasive electrodes on the neck or auricle for stimulation of the cervical or auricular branch of the vagus nerve respectively(7). Transcutaneous VNS has a lower risk of adverse events, is reversible and easy to implement(7). In addition, experimental evidence suggests that the effects of transcutaneous VNS on brain function are comparable to those obtained with VNS(8).

This study will evaluate the effects of transcutaneous vagus nerve stimulation (tVNS) in combination with physical rehabilitation on upper limb motor function of patients with stroke. Thirty patients with ischemic stroke will be included in the study. Subjects will be randomized to tVNS + physical rehabilitation or sham stimulation + physical rehabilitation. Therapy sessions will be performed 3 times a week for six consecutive weeks. Efficacy will be evaluated by assessing the change in motor function of the upper limb, the next day and 30 days after the end of the intervention. The motor function of the upper limb will be assessed by means of the Fugl-Meyer scale score.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <75 years
* Unilateral supratentorial ischemic stroke that occurred at least 7 days but not more 30 days before enrollment.
* Modified Rankin Scale between 0 and 1 before stroke
* Contralesional UL motor impairment defined by NIHSS item 5 score ≥ 1 to ≤ 3.
* Ability to provide written informed consent.
* Hemodynamically stable patients.
* Patients residing in the metropolitan area of Bucaramanga.

Exclusion Criteria:

* Significant cognitive or language impairment that would interfere with study participation or informed consent. This criterion will be defined by NIHSS item 1a-c score > 2, item 9 score > 1, item 11 score = 2.
* Medical conditions that could interfere with study participation, for example ear infections or skin wounds.
* Bradycardia (< 50 bpm) or hypotension (< 90/60 mmHg)
* Significant pre-existing disability
* History of stroke
* History of cardiac arrhythmia
* History of severe head trauma, brain surgery, deep brain stimulation, or brain injuries of other etiologies.
* Pregnant or planning on becoming pregnant or breastfeeding during the study period.
* Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse) that would prevent subject from meeting protocol timeline.
* Subjects who are currently in another clinical trial or plan to do so during the study period.
* Patient receiving any therapy at study entry that would interfere with VNS (e.g., drugs that interfere with neurotransmitter mechanisms: anticholinergics, adrenergic blockers, etc.).
* Prior injury to vagus nerve.
* Any other implanted device such as a pacemaker or other neurostimulator; any other investigational device or drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Motor function of the upper limb | 1 day and 30 days after the end of the intervention
  Efficacy will be assessed by evaluating the change in motor function of the upper limb, the next day and 30 days after the end of the intervention. The motor function of the upper limb will be assessed by means of the Fugl-Meyer scale score. The motor function component ranges from 0 to 100, where higher scores indicate better motor recovery.
Arm and hand mobility Description: | 1 day and 30 days after the end of the intervention
  Change in arm mobility the next day and 30 days after the end of the intervention. Arm and hand mobility will be assessed by the ARAT test. The maximum score on the ARAT is 57 points ( 0 to 57). A higher score indicates better arm function.

SECONDARY OUTCOMES:
Hospital anxiety and depression | 1 day and 30 days after the end of the intervention
  Change in anxiety and depression symptoms the next day and 30 days after the end of the intervention. The anxiety and depression symptoms will be assessed by means of the HADS scale score. Each subscale score ranges from 0 to 21, and higher scores indicate more severe anxiety and/or depressive symptoms.
Medical device safety | During the intervention period.
  Adverse events associated with the stimulation, device and health attention are associated. It would be a measure of the number of events related or not related to the device. Each adverse event should be asses by ethical committee and medical team.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Sanabria, Bacteriologist, PhD, Study Director — Fundación Cardiovascular de Colombia
Locations (1):
- Neurology Center of Excellence - Hospital Internacional de Colombia - Fundación cardiovascular de Colombia, Piedecuesta, Santander Department, Colombia

REFERENCES:
- [Background] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part II. Headache. 2016 Feb;56(2):259-66. doi: 10.1111/head.12650. Epub 2015 Sep 18. PMID 26381725
- [Background] Yap JYY, Keatch C, Lambert E, Woods W, Stoddart PR, Kameneva T. Critical Review of Transcutaneous Vagus Nerve Stimulation: Challenges for Translation to Clinical Practice. Front Neurosci. 2020 Apr 28;14:284. doi: 10.3389/fnins.2020.00284. eCollection 2020. PMID 32410932
- [Background] van der Meij A, Wermer MJH. Vagus nerve stimulation: a potential new treatment for ischaemic stroke. Lancet. 2021 Apr 24;397(10284):1520-1521. doi: 10.1016/S0140-6736(21)00667-X. No abstract available. PMID 33894818
- [Background] Kong KH, Chua KS, Lee J. Recovery of upper limb dexterity in patients more than 1 year after stroke: Frequency, clinical correlates and predictors. NeuroRehabilitation. 2011;28(2):105-11. doi: 10.3233/NRE-2011-0639. PMID 21447911
- [Background] Dancause N, Nudo RJ. Shaping plasticity to enhance recovery after injury. Prog Brain Res. 2011;192:273-95. doi: 10.1016/B978-0-444-53355-5.00015-4. PMID 21763529
- [Background] Cramer SC. Repairing the human brain after stroke: I. Mechanisms of spontaneous recovery. Ann Neurol. 2008 Mar;63(3):272-87. doi: 10.1002/ana.21393. PMID 18383072
- [Background] Nakayama H, Jorgensen HS, Raaschou HO, Olsen TS. Recovery of upper extremity function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1994 Apr;75(4):394-8. doi: 10.1016/0003-9993(94)90161-9. PMID 8172497
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265